CLINICAL TRIAL: NCT07124117
Title: A Phase 1/2, Open-Label, Dose-Escalation and Cohort-Expansion Study Evaluating the Safety, Pharmacokinetics, and Therapeutic Activity of OBI-902 in Participants With Advanced Solid Tumors
Brief Title: A Study Evaluating OBI-902 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OBI-902-001
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Phase 1a Dose Escalation: Cohort 1 (Experimental): OBI-902 at dose level 1.6 mg/kg, Q3W
  Interventions: Drug: OBI-902
- Phase 1a Dose Escalation: Cohort 2 (Experimental): OBI-902 at dose level 3.0 mg/kg, Q3W
  Interventions: Drug: OBI-902
- Phase 1a Dose Escalation: Cohort 3 (Experimental): OBI-902 at dose level 4.5 mg/kg, Q3W
  Interventions: Drug: OBI-902
- Phase 1a Dose Escalation: Cohort 4 (Experimental): OBI-902 at dose level 6.0 mg/kg, Q3W
  Interventions: Drug: OBI-902
- Phase 1a Dose Escalation: Cohort 5 (Experimental): OBI-902 at dose level 8.0 mg/kg, Q3W
  Interventions: Drug: OBI-902
- Phase 1a Dose Escalation: Cohort 6 (Experimental): OBI-902 at dose level 10.0 mg/kg, Q3W
  Interventions: Drug: OBI-902
- Phase 1b Cohort Expansion: Cohort 1 (Experimental): OBI-902 at the putative RP2D determined during the Phase 1a Dose Escalation; biliary tract cancer cohort.
  Interventions: Drug: OBI-902
- Phase 1b Cohort Expansion: Cohort 2 (Experimental): OBI-902 at the putative RP2D determined during the Phase 1a Dose Escalation; gastric and gastroesophageal cancer cohort.
  Interventions: Drug: OBI-902
- Phase 1b Cohort Expansion: Cohort 3 (Experimental): OBI-902 at the putative RP2D determined during the Phase 1a Dose Escalation; platinum resistant ovarian cancer cohort.
  Interventions: Drug: OBI-902
- Phase 2 Randomized Dose Optimization Cohort: Cohort 1 (Experimental): Randomized dose optimization cohort. Tumor type and/or population will be based on safety/tolerability, PK, and preliminary efficacy of OBI-902 from Phase 1 part of the study.
  Interventions: Drug: OBI-902
- Phase 2 Randomized Dose Optimization Cohort: Cohort 2 (Experimental): Randomized dose optimization cohort. Tumor type and/or population will be based on safety/tolerability, PK, and preliminary efficacy of OBI-902 from Phase 1 part of the study.
  Interventions: Drug: OBI-902

INTERVENTIONS:
Drug: OBI-902 — OBI-902 is an antibody-drug conjugate study drug

SUMMARY:
This is a 3-part study. Phase 1a (dose escalation) is designed to assess the safety and tolerability and to determine the maximum tolerated dose (MTD) and putative recommended phase 2 dose (RP2D) of study drug as monotherapy. Phase 1b (Cohort Expansion) is intended to further characterize the safety and preliminary antitumor activity of the putative RP2D of OBI-902 in selected tumor types. Phase 2 (Randomized Dose Optimization Cohorts) is intended to determine the optimal RP2D of OBI-902 in selected tumor types, before advancing to larger Phase 3 trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, 18 years of age or older at the time of consent
2. Provide written informed consent prior to performing any study-related procedure
3. Histologically or cytologically confirmed participants with metastatic or advanced solid tumor that is not curable with local therapies
4. Participants must have been treated with established standard-of-care therapy, andphysicians have determined that such established therapy is not sufficiently efficacious, or patients have declined to receive standard-of-care therapy. In the latter case, the source documentation must state the effective therapies the participant is declining.
5. Measurable disease (i.e., at least one measurable lesion per RECIST 1.1)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Adequate organ function defined as:

   a. Hepatic:

   i. Serum ALT ≤3 × upper limit of normal (ULN), ≤5 × ULN in the presence of liver metastases

   i. Serum AST ≤3 × ULN, ≤5 × ULN in presence of liver metastases

   ii. Serum bilirubin ≤1.5 × ULN (unless due to Gilbert's syndrome (typically elevated total bilirubin of 1-5 mg/dL with a normal direct bilirubin) or hemolysis)

   b. Creatinine clearance >60 mL/minute using Modification of Diet in Renal Disease equation

   c. Hematologic:

   i. ANC ≥1,500/µL (>1,200/µL in Duffy antigen-null participants)

   ii. Platelets ≥100,000/µL

   iii. Hemoglobin ≥8 g/dL
8. Participants must be willing and able to comply with all protocol-required assessments, visits, and procedures, including evaluable pretreatment tumor biopsy. Archival tumor biopsies are acceptable at baseline.
9. Females of childbearing potential must have negative serum pregnancy test prior to starting study therapy and agree to use a reliable form of contraceptive during the study treatment period and for at least 7 months following the last dose of study drug.
10. Participants not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in the trial. Postmenopausal is defined as 12 months with no menses without an alternative medical cause. Male participants must agree to use an adequate method of contraception during the study treatment period and for at least 4 months following the last dose of study drug.
11. Participants with human immunodeficiency virus (HIV) infection or with documented history of HIV infection are eligible if CD4+ T-cell counts are ≥350 cells/μL and have an HIV viral load less than 200 copies/mL prior to enrollment. Participants on ART should be on an established dose for at least 4 weeks under stable condition.
12. Participants with serological evidence of chronic HBV infection or with documented history of HBV infection are eligible if they have an HBV viral load below the limit of quantification with or without concurrent viral suppressive therapy.
13. Participants with a history of HCV infection can be under curative antiviral treatment and have a viral load below the limit of quantification.
14. Participants in Phase 1b (Cohort Expansion) - must have one of the following tumor types to be enrolled in the respective cohort:

    * Cohort 1: BTC (intra- and extrahepatic CCA, carcinoma of ampulla of Vater, and gallbladder disease)
    * Cohort 2: Gastric and GEJ cancer
    * Cohort 3: PROC

Exclusion Criteria:

1. Less than 3 weeks from prior cytotoxic chemotherapy or radiation therapy; and less than 5 half-lives or 3 weeks, whichever is shorter, from prior biologic therapies, prior to the first dose of OBI-902.
2. Participants that have undergone a major surgical procedure (as defined by the investigator) or significant traumatic injury within 28 days prior to the first dose of OBI-902.
3. Sensory or motor neuropathy of Grade 2 or greater.
4. Participants with a history of solid organ transplants. Corneal transplant without immunosuppressive therapy is allowed.
5. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using NCI CTCAE version 5.0), except for alopecia and laboratory values listed in the inclusion criteria.
6. Receipt of any prior therapy targeting TROP2. (Phase 2 only)
7. Corrected QT interval (QTcF) prolongation to >470 msec based on the average of the screening 12-lead ECGs
8. Known hypersensitivity to OBI-902 or its excipients.
9. Participants with known untreated central nervous system (CNS) metastases. Participants with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period.
10. Participants with significant clinical cardiac abnormality (e.g., clinical heart failure or unstable angina).
11. Any medical comorbidity that is life-threatening or, in the opinion of the Investigator, renders the participant unsuitable for participation in a clinical trial due to possible noncompliance, would place the participant at an unacceptable risk and/or potential to affect interpretation of results of the study.
12. Participants who are pregnant or breastfeeding.
13. Is receiving any concurrent prohibited medications as listed in OBI-902-001 clinical protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-02-08 (Estimated); Study Completion 2029-02-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of OBI-902: incidence of adverse events (AEs) and serious adverse events (SAEs), changes in selected clinical laboratory parameters, cardiac parameters, and vital signs. | Duration of study, up to 54 weeks
  To assess the safety and tolerability of OBI-902 when administered intravenously to participants with advanced solid tumors
Maximum tolerated dose (MTD) of OBI-902 | Duration of study, up to 54 weeks
  To determine the MTD of OBI-902 at which the pre-defined rate of dose limiting toxicities (DLTs) is not exceeded.
Preliminary antitumor activity of OBI-902 in selected tumor types - Objective Response Rate (ORR) | Duration of study, up to 54 weeks
  Percentage of participants with ORR according to RECIST version 1.1 for each cohort
Preliminary antitumor activity of OBI-902 in selected tumor types - Duration of Response (DoR) | Duration of study, up to 54 weeks
  Percentage of participants with DOR according to RECIST version 1.1 for each cohort
Preliminary antitumor activity of OBI-902 in selected tumor types - Clinical Benefit Rate (CBR) | Duration of study, up to 54 weeks
  Percentage of participants with CBR according to RECIST version 1.1 for each cohort
Preliminary antitumor activity of OBI-902 in selected tumor types - Disease Control Rate (DCR) | Duration of study, up to 54 weeks
  Percentage of participants with DCR according to RECIST version 1.1 for each cohort
Safety and tolerability of OBI-902 in Phase 1b/Phase 2: incidence of AEs, SAEs, and laboratory abnormalities. | Duration of study, up to 54 weeks
  To further characterize safety and tolerability of OBI-902 as graded by NCI CTCAE version 5.0.
Optimal recommended phase 2 dose (RP2D) of OBI-902 | Duration of study, up to 54 weeks
  To determine the optimal RP2D of OBI-902 for larger Phase 3 trials

SECONDARY OUTCOMES:
Preliminary long-term efficacy of OBI-902 in selected tumor types | Duration of study, up to 54 weeks
  PFS as assessed by the investigator and OS.
Pharmacokinetics (PK) of OBI-902 and exatecan: Peak Plasma Concentration (Cmax) | Duration of study, up to 54 weeks
  To evaluate the serum Cmax of OBI-902 and exatecan
Pharmacokinetics (PK) of OBI-902 and exatecan: area under the concentration-time curve (AUC) | Duration of study, up to 54 weeks
  To evaluate the serum AUC of OBI-902 and exatecan
Pharmacokinetics (PK) of OBI-902 and exatecan: half-life (T1/2) | Duration of study, up to 54 weeks
  To evaluate the serum half-life of OBI-902 and exatecan
Pharmacokinetics (PK) of OBI-902 and exatecan: clearance (CL) | Duration of study, up to 54 weeks
  To evaluate the serum clearance of OBI-902 and exatecan
Pharmacokinetics (PK) of OBI-902 and exatecan: volume distribution at steady state (Vdss) | Duration of study, up to 54 weeks
  To evaluate the serum volume distribution at steady state of OBI-902 and exatecan
Immunogenicity of OBI-902 | Duration of study, up to 54 weeks
  To evaluate the immunogenicity of OBI-902 anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Scripps Green Hospital, La Jolla, California
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Taiwan (3):
  - Wan Fan Hospital, Taipei, Wenshan
  - Shuang Ho Hospital, Taipei, Zhonghe
  - China Medical University Hospital, Taichung